CLINICAL TRIAL: NCT06075979
Title: The First Affiliated Hospital of Shandong First Medical University
Brief Title: Correlation Between Microbial Infection and Lumbar Degenerative Disease Based on High-throughput Gene Sequencing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HaoxuanZhang (Other)
Responsible Party: Sponsor-Investigator, HaoxuanZhang, Associate professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Other
Other Study IDs: High-throughput gene
Record Dates: First submitted 2023-09-18; First posted 2023-10-10 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Lumbar Degenerative Diseases; Gene Product Sequence Variation
Keywords: lumbar degenerative diseases; high-throughput gene sequencing; microbial infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbar disc herniation group (Experimental): Patients undergoing surgery for lumbar disc herniation
  Interventions: Other: Lumbar disc herniation; Other: Lumbar spinal stenosis
- Lumbar spinal stenosis group (Experimental): Patients undergoing surgery for lumbar spinal stenosis
  Interventions: Other: Lumbar disc herniation; Other: Lumbar spinal stenosis

INTERVENTIONS:
Other: Lumbar disc herniation — Patients undergoing surgery for lumbar disc herniation
Other: Lumbar spinal stenosis — Patients undergoing surgery for lumbar spinal stenosis

SUMMARY:
Lumbar degenerative disease is one of the most common diseases in orthopedic and spinal surgery. The pathogenesis of lumbar degenerative disease is still unclear, mainly including aging degeneration and biomechanical hypothesis. In our previous research work，the investigators took lumbar disc tissue from patients who underthe investigatorsnt surgical treatment for lumbar degenerative diseases. The investigators found that some patients had low-toxic bacterial infection in the intervertebral disc tissue. Combined with literature and previous studies, it is suggested that microbial infection plays a role in lumbar degenerative diseases. The investigators suggest that microbial infection may be closely related to the occurrence and development of lumbar degenerative diseases, which may cause or even accelerate the degeneration of lumbar intervertebral disc tissue. The current research difficulties are as follows: 1. Low sensitivity and specificity of microbial analysis; 2. It is difficult to distinguish the colonization infection of intervertebral disc tissue microorganisms from the contamination of foreign substances. In view of this, this study intends to use the high-throughput gene sequencing technology of infectious pathogens based on nano single molecule sequencing, double verification of blood samples and intervertebral disc tissue samples, to identify the microbial status of degenerative lumbar disc tissue, and to explore the correlation between lumbar degenerative disease and microbial infection, identifying relevant susceptible microorganisms, which is expected to study the pathogenesis of this susceptible microorganism in the future, and provide new ideas and approaches for the prevention, control and treatment of lumbar degenerative diseases.

DETAILED DESCRIPTION:
This study intends to use the high-throughput gene sequencing technology of infectious pathogens based on nano single molecule sequencing, double verification of blood samples and intervertebral disc tissue samples, to identify the microbial status of degenerative lumbar disc tissue, and to explore the correlation between lumbar degenerative disease and microbial infection, identifying relevant susceptible microorganisms, which is expected to study the pathogenesis of this susceptible microorganism in the future, and provide new ideas and approaches for the prevention, control and treatment of lumbar degenerative diseases.This clinical study has a funding of 50000 RMB.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the experimental group, aged 18 to 85 years old, have symptoms and imaging data that support the diagnosis of lumbar degenerative diseases (including lumbar disc herniation, lumbar spinal stenosis, and lumbar spondylolisthesis).
* Patients who undergo strict conservative treatment for 3 months before surgery have no significant improvement in symptoms; The control group of patients had no significant lumbar disc degeneration evaluated by imaging, but needed surgical decompression and fusion intervention due to trauma causing lumbar fractures, lumbar tumors, scoliosis.
* The disc organizer can be obtained during surgery.

Exclusion Criteria:

* Lumbar degenerative diseases combined with infectious diseases.
* Lumbar degenerative diseases combined with mental diseases.
* Lumbar degenerative diseases combined with metal allergy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Classification of endplate degeneration in lumbar magnetic resonance imaging - Modic classification | 3 years
  Modic degeneration of the vertebral endplate in the lumbar spine refers to a common abnormal signal change in the endplate and subendplate bone on lumbar magnetic resonance imaging after excluding tumors and tuberculosis. It reflects the microscopic changes in tissue biochemistry within the endplate and the manifestations of endplate degeneration. Modic and other scholars have conducted detailed research on it and classified it into three types based on the signal level and pathological and biochemical changes on MRI, as shown in Figure 1. Type I (edema type): Low signal on T1WI, high signal on T2WI, and cracks in the endplate can be found in the granulation tissue of new blood vessels in the bone marrow; Type II (fatty type): High signal on T1WI, equal or slightly high signal on T2WI, adjacent bone marrow tissue replaced by adipocytes, and end plate rupture; Type III (sclerotic type): Low signal on T1WI and T2WI, with sclerosis changes in the endplate and subchondral bone.
Classification of intervertebral disc degeneration -Pfirrmann classification | 3 years
  The Pfirmmann grading system based on sagittal T2WI of lumbar magnetic resonance imaging is a semi quantitative evaluation method for the degree of lumbar disc degeneration, which can display the morphological changes of lumbar disc degeneration. It is currently a widely used and highly recognized grading system for evaluating the degree of lumbar disc degeneration. This grading system was proposed by Pfirmmann in 2001, which evaluates the level of lumbar disc degeneration based on indicators such as signal intensity, disc shape, and intervertebral space changes in the midsagittal position of the T2WI sequence.
General bacterial culture and identification | 3 years
  Collect blood samples from patients before surgery and intervertebral disc tissue after decompression during surgery. Send blood samples and intervertebral disc tissue samples to bacterial culture analysis for microbial species and drug sensitivity, and conduct smear observation, aerobic and anaerobic environment culture identification. The VitekII Compact fully automated microbial identification and drug sensitivity analysis system (BioMerieux, Marcy Ioile, France) was used for bacterial identification and sensitivity testing of commonly used clinical drugs, and the paper diffusion method (K-B method) was used to increase sensitivity testing of commonly used antibiotics such as levofloxacin, polymyxin B, cefoperazone/sulbactam, minocycline, and vancomycin.
High throughput gene sequencing and drug sensitivity analysis of infectious pathogens | 3 years
  Collect blood samples from patients before surgery, and collect intervertebral disc tissue from patients after decompression during surgery using sterile collection tubes. To ensure the comprehensive identification of microbial species, this study plans to simultaneously sequence RNA and DNA using the TIAAmp MicroRNA and DNA Extraction Kit (Beijing Tiangen Biochemical Technology Co., Ltd., China), and extract RNA and DNA from blood samples and intervertebral disc tissue samples according to the instructions in the manual.
  For microbial data analysis, use the Sanger method to map the sequencing results in BWA; Convert data to bam format using SAMtools; After using the built-in script of the software for filtering, use IGV software to process the mapping data; Assemble consistent sequences using SAMTools and BCFtools; Visualize using IGV software; Verify the sequencing accuracy of Nanopore MinION by comparing consistent sequences and Sanger method reference sequences.

SECONDARY OUTCOMES:
VAS | 3 years
  The visual analog scale (VAS) is used for pain assessment. It is widely used in clinical practice in China, and the basic method is to use a vernier ruler with a length of about 10cm, marked with 10 scales on one side, with both ends marked as "0" and "10" respectively. A score of 0 indicates painlessness, and a score of 10 represents the most severe pain that cannot be tolerated.
JOA | 3 years
  The Japanese Orthopaedic Association Scores (JOA) is a neurological function scoring system recommended by the Japanese Orthopaedic Association, which includes four parts: upper limb motor function, lower limb motor function, sensory and bladder function, with a total score of 29 points. The lower the score, the more severe the neurological dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Hao-Xuan Zhang, Ph.D/MD, Study Chair — Shandong First Medical University
Locations (1):
- Hao-Xuan Zhang, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No